CLINICAL TRIAL: NCT05973474
Title: Prognostic Value of the Atherogenic Index of Plasma（AIP）for Cardiovascular Outcomes in Patients With Atrial Fibrillation
Brief Title: The Atherogenic Index of Plasma（AIP） in Patients With Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, zhangkun, associate chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-634-01
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Atrium; Fibrillation; Lipid Metabolism Disorders; Cardiovascular Diseases; Event, Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Lipid Metabolism Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about The Atherogenic Index of Plasma(AIP) in patients with atrial fibrillation(AF). The main questions it aims to answer are: (1)To investigate the correlation between AIP and the occurrence rate of AF. (2) To investigate the correlation between AIP and the occurrence rate of cardiovascular outcome events (MACE events, heart failure, embolism events) in patients with AF. Patients's clinical data including medical history, laboratory tests, and imageological examination will be collected and further analysed.

DETAILED DESCRIPTION:
Baseline demographic data: age, gender, height, weight, systolic blood pressure, diastolic blood pressure, smoking habit, drinking habit, physical activity, fasting blood glucose, medication use (statins, ACEI/ARB, anticoagulant related drugs), basic medical history (hypertension, diabetes mellitus, coronary heart disease).

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation was detected by electrocardiogram or 24-hour holter or portable electrocardiogram monitor;
2. age ≥18 years old;
3. "low-intermediate" risk group of AF cardioembolic stroke: male patients with CHA2DS2-VASc score 0-1 or female patients with CHA2DS2-VASc score 1-2

Exclusion Criteria:

1. patients with rheumatic heart disease, congenital heart disease, cardiomyopathy, hematological diseases, severe hepatic and renal insufficiency and connective tissue diseases;
2. Echocardiography showed valvular heart disease;
3. patients with transient atrial fibrillation secondary to reversible causes: hyperthyroidism, acute pulmonary embolism, recent surgery, acute myocardial infarction, etc.
4. severe carotid artery stenosis and intracranial artery stenosis;
5. AF patients with recent major surgery.
6. patients with serious lack of clinical data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with AF during hospitalization in our hospital.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation (AF) | 10 years
  AF diagnoses were ascertained by 3 different sources in our study: ECGs performed at study visits, hospital discharge codes, and death certificates. All ECGs automatically coded as AF were visually checked by a trained cardiologist to confirm AF diagnosis.

SECONDARY OUTCOMES:
major adverse cardiovascular events (MACEs) | 10 years
  Follow up main adverse cardiovascular and cerebrovascular events such as death, myocardial infarction, stroke, and repeated revascularization.
heart failure | 10 years
  Patients who required intravenous medications for heart failure after admission (including diuretics, vasodilators, or inotropic agents) or a significant increase in the dose of oral diuretics (i.e., an increase in furosemide of ≥40mg or equivalent or the addition of a thiazide to a loop diuretic) were considered to have heart failure readmission. Pulmonary rales and/or the third heart sound, chest X-ray, dyspnea, peripheral edema, and NYHA grade were evaluated to further confirm the occurrence of heart failure.